CLINICAL TRIAL: NCT01525589
Title: A Multicenter Phase II Clinical Trial of PM01183 in BRCA 1/2-Associated or Unselected Metastatic Breast Cancer
Brief Title: A Phase II Clinical Trial of PM01183 in BRCA 1/2-Associated or Unselected Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-B-003-11
Record Dates: First submitted 2012-01-30; First posted 2012-02-03 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; PM01183; lurbinectedin; Pharma Mar
MeSH Terms: conditions — Breast Neoplasms | interventions — PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PM01183 (Experimental)
  Interventions: Drug: PM01183

INTERVENTIONS:
Drug: PM01183 — PM01183 drug product (DP) is presented as a lyophilized powder for concentrate for solution for infusion with two strengths: 1 mg/vial and 4 mg/vial

SUMMARY:
A Clinical Trial of PM01183 in Metastatic Breast Cancer to assess the antitumor activity of PM01183 ,to evaluate whether the presence of a known germline mutation in BRCA 1/2 predicts response to PM01183 in Metastatic Breast Cancer (MBC) patients, to evaluate the safety profile of this PM01183 to analyze the pharmacokinetics (PK) and PK/PD (pharmacokinetic/pharmacodynamic) correlations and to evaluate the pharmacogenomic (PGx) expression profile in tumor samples.

DETAILED DESCRIPTION:
A Multicenter Phase II Clinical Trial of PM01183 in BRCA 1/2-Associated or Unselected Metastatic Breast Cancer to assess the antitumor activity of PM01183 in terms of overall response rate (ORR), duration of response (DR),clinical benefit [ORR or stable disease lasting over three months (SD > 3 months)], progression free survival (PFS), and one-year overall survival (1y-OS) and to evaluate whether the presence of a known germline mutation in BRCA 1/2 predicts response to PM01183 in MBC patients, to explore the activity of PM01183 in specific breast cancer subpopulations according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications, to evaluate the safety profile of this PM01183 administration schedule [Day 1 every three weeks (q3wk)] in this patient population, to analyze the pharmacokinetics (PK) of PM01183 in this patient population, to explore PK/PD (pharmacokinetic/ pharmacodynamic) correlations, if applicable and to evaluate the pharmacogenomic (PGx) expression profile of selected putative markers potentially predictive of response to PM01183, in tissues from tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 and ≤ 75 years of age.
* Voluntary signed informed consent form (ICF).
* Proven diagnosis of metastatic breast cancer (MBC).
* At least one, but no more than three, prior chemotherapy regimens for MBC.
* Patients with known HER-2 overexpressing MBC must have failed at least one prior trastuzumab-containing regimen for metastatic disease.
* Disease evaluable for response by specific appropriate criteria.
* No or minimal disease-related symptoms not affecting patient daily activities.
* Adequate major organ function (normal or minimal alteration in liver, kidney, hematological, metabolic and cardiac function)
* Wash out periods prior to Day 1 of Cycle 1:

At least three weeks since the last chemotherapy (six weeks in some particular cases) and At least four weeks since the last radiotherapy (RT) > 30 Gy) and At least one week since the last hormonal therapy and At least two weeks since the last biological/investigational therapy

* Minimal or no ongoing toxicity from immediately prior therapy according to specific appropriate criteria. Mild ongoing toxicity is allowed in case of alopecia, skin toxicity, fatigue and/or finger numbness or tumbling.
* Patients of child-bearing potential must agree to use a medically approved contraception method until at least six weeks after the last study drug administration.
* Known deleterious germline mutation of BRCA1/2 (Patients in Cohorts A and A1)
* Prior treatment with PARP inhibitors (Patients in Cohort A1)

Exclusion Criteria:

* Prior treatment with PM01183 or trabectedin.
* Extensive prior RT.
* Prior or concurrent malignant disease unless cured for more than five years.
* Exceptions are breast cancer in the other breast.
* Uncommon or rare subtypes of breast cancer.
* Symptomatic or progressive brain metastases.
* Bone-limited and exclusively metastases.
* Relevant diseases or clinical situations which may increase patient's risk:

History of cardiac disease. Moderate breathing difficulties or oxygen requirement Active uncontrolled infection. Unhealed wound or presence of any external drainage. Chronically active viral hepatitis. Immunocompromised patients, including those known to be infected by human immunodeficiency virus (HIV).

Known muscular disease or functional alteration

* Pregnant or breastfeeding women.
* Impending need for immediate RT for symptomatic relief.
* Limitation of the patient's ability to comply with the treatment or to follow-up the protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Stanford Women's Cancer Center, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Abramson Cancer Center - Hospital of the University of Pennsylvania at Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (4):
  - Complexo Hospitalario Universitario A Coruña, A Coruña, A Coruña
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Fernandez-Teruel C, Lubomirov R, Fudio S. Population Pharmacokinetic-Pharmacodynamic Modeling and Covariate Analyses of Neutropenia and Thrombocytopenia in Patients With Solid Tumors Treated With Lurbinectedin. J Clin Pharmacol. 2021 Sep;61(9):1206-1219. doi: 10.1002/jcph.1886. Epub 2021 Jun 9. PMID 33914350
- [Derived] Cruz C, Llop-Guevara A, Garber JE, Arun BK, Perez Fidalgo JA, Lluch A, Telli ML, Fernandez C, Kahatt C, Galmarini CM, Soto-Matos A, Alfaro V, Perez de la Haza A, Domchek SM, Antolin S, Vahdat L, Tung NM, Lopez R, Arribas J, Vivancos A, Baselga J, Serra V, Balmana J, Isakoff SJ. Multicenter Phase II Study of Lurbinectedin in BRCA-Mutated and Unselected Metastatic Advanced Breast Cancer and Biomarker Assessment Substudy. J Clin Oncol. 2018 Nov 1;36(31):3134-3143. doi: 10.1200/JCO.2018.78.6558. Epub 2018 Sep 21. PMID 30240327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was included on 27JUN12 and the first study treatment administration was on 28JUN12.
  The cutoff date for the results was 24OCT18. A total of 111 patients were included in the 3 cohorts of the study: 56 in Cohort A (BRCA+), 20 in Cohort A1 (BRCA+/PARPi), 35 in Cohort B (Unselected).
Groups:
- Cohort A (BRCA+): Patients with known deleterious BRCA1/2 mutation status at study entry
- Cohort A1 (BRCA+/PARPi): Patients with known deleterious BRCA1/2 mutation status and prior treatment with PARPi.
- Cohort B (Unselected): Patients without known deleterious BRCA1/2 mutation status at study entry, i.e., either:
  * Patients known to have no deleterious BRCA1/2 mutations (BRCA-), or
  * Patients whose BRCA 1/2 mutation status was unknown (BRCA-UK). BRCA1/2 germline mutation status would be assessed in all patients in this subgroup responding to lurbinectedin treatment.
Period: Overall Study
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Started | 56 | 20 | 35
Completed | 0 | 0 | 0
Not Completed | 56 | 20 | 35
Not completed — Non-treatment-related AE | 1 | 0 | 0
Not completed — Progressive disease | 48 | 15 | 29
Not completed — Never treated | 2 | 0 | 0
Not completed — Physician Decision | 4 | 2 | 2
Not completed — Death | 0 | 0 | 2
Not completed — Treatment-related AE | 1 | 1 | 2
Not completed — Other reasons | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected) | Total
Number analyzed (Participants) | 56 | 20 | 35 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 19 | 30 | 100
  >=65 years | 5 | 1 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 42.5 [30 to 73] | 45.0 [31 to 66] | 52.0 [32 to 70] | 45.0 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 20 | 35 | 111
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 50 | 16 | 32 | 98
  Race: Black | 2 | 0 | 1 | 3
  Race: Asian | 1 | 1 | 0 | 2
  Race: Hispanic | 2 | 1 | 2 | 5
  Race: Unknown | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 16 | 9 | 60
  Spain | 21 | 4 | 26 | 51
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active, able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours PS 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours PS 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 32 | 10 | 22 | 64
    PS 1 | 24 | 10 | 13 | 47
Sites of disease at diagnosis [Count of Participants; unit: Participants]
  Left breast | 26 | 11 | 18 | 55
  Right breast | 28 | 9 | 15 | 52
  Bilateral | 2 | 0 | 2 | 4
Histology type at diagnosis [Count of Participants; unit: Participants]
  Ductal carcinoma | 54 | 20 | 34 | 108
  Lobular carcinoma | 2 | 0 | 0 | 2
  Lobular and ductal carcinoma | 0 | 0 | 1 | 1
Histology grade at diagnosis [Count of Participants; unit: Participants] — Well differentiated: The cells are slower-growing, and look more like normal breast tissue.
  Moderately differentiated: The cells are growing at a speed of and look like cells somewhere between grades 1 and 3.
  Poorly differentiated: The cancer cells look very different from normal cells and will probably grow and spread faster.
  Participants
    Well differentiated | 3 | 0 | 1 | 4
    Moderately differentiated | 10 | 8 | 13 | 31
    Poorly differentiated | 31 | 11 | 17 | 59
    Unknown | 12 | 1 | 4 | 17
Stage at diagnosis [Count of Participants; unit: Participants] — Stage I describes invasive breast cancer (cancer cells are breaking through to or invading normal surrounding breast tissue) Stage II. The cancer has grown, spread, or both. Stage III. The cancer has not spread to bones or organs, but it's considered advanced, and it's harder to fight.
  Stage IV describes invasive breast cancer that has spread beyond the breast and nearby lymph nodes to other organs of the body, such as the lungs, distant lymph nodes, skin, bones, liver, or brain.
  Participants
    Stage I | 9 | 3 | 0 | 12
    Stage II | 26 | 9 | 13 | 48
    Stage III | 16 | 6 | 19 | 41
    Stage IV | 5 | 2 | 3 | 10
BRCA deleterious mutation [Count of Participants; unit: Participants]
  BRCA1 | 33 | 10 | 0 | 43
  BRCA2 | 23 | 9 | 0 | 32
  Both | 0 | 1 | 0 | 1
  Not applicable | 0 | 0 | 35 | 35
Hormonal status [Count of Participants; unit: Participants]
  Triple negative | 33 | 7 | 17 | 57
  ER and/or PR positive and HER2 negative | 21 | 12 | 14 | 47
  ER and/or PR positive and HER2 positive | 2 | 1 | 3 | 6
  ER and PR negative and HER2 positive | 0 | 0 | 1 | 1
Sites at baseline [Count of Participants; unit: Participants]
  <3 sites | 23 | 7 | 21 | 51
  ≥3 sites | 33 | 13 | 14 | 60
Prior surgery [Count of Participants; unit: Participants] | 53 | 19 | 34 | 106
Prior radiotherapy [Count of Participants; unit: Participants] | 44 | 18 | 32 | 94
Weight [Median (Full Range); unit: Kg] | 69.2 [48.4 to 107.3] | 59.8 [48.5 to 98.8] | 71.7 [43.0 to 153.6] | 68.1 [43.0 to 153.6]
Height [Median (Full Range); unit: cm] | 162.5 [150.0 to 178.0] | 161.0 [148.0 to 173.0] | 161.0 [147.0 to 171.0] | 162.0 [147.0 to 178.0]
Body Surface Area [Median (Full Range); unit: m^2] | 1.72 [1.47 to 2.12] | 1.63 [1.48 to 2.05] | 1.75 [1.36 to 2.41] | 1.72 [1.36 to 2.41]
Albumin [Median (Full Range); unit: g/dL] | 4.1 [3.3 to 4.9] | 4.1 [3.6 to 4.8] | 4.0 [3.4 to 4.6] | 4.1 [3.3 to 4.9]
Number of sites at baseline [Median (Full Range); unit: sites] | 3.0 [1 to 7] | 3.0 [1 to 6] | 2.0 [1 to 6] | 3.0 [1 to 7]
Time from first diagnosis to registration [Median (Full Range); unit: months] | 44.0 [0.9 to 170.3] | 55.7 [11.5 to 337.3] | 47.0 [5.0 to 177.3] | 46.5 [0.9 to 337.3]
Time from metastatic disease to registration [Median (Full Range); unit: months] | 12.5 [0.4 to 129.8] | 26.1 [8.4 to 98.2] | 13.8 [2.5 to 110.9] | 14.8 [0.4 to 129.8]
Time from last progression before study entry [Median (Full Range); unit: weeks] | 2.9 [0 to 15.6] | 3.2 [0.9 to 14.0] | 3.0 [0.7 to 8.1] | 3.0 [0.0 to 15.6]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The overall response rate is defined as the percentage of patients with a confirmed response, either complete response (CR) or partial response (PR), according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1. Per RECIST v1.1 for target lesions and assessed by MRI: CR, Disappearance of all target lesions; PR >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Minimum 10-12 months if negative results and up to 26-28 months if study is to be complete the targeted enrollment
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage | 40.7 [27.6 to 55.0] | 5.0 [0.1 to 24.9] | 8.8 [1.9 to 23.7]

2. Primary Outcome: Overall Response
Description: Overall Response Rate (ORR) in the population evaluable for efficacy according to RECIST v.1.1. ORR was defined as the percentage of patients with a confirmed response, either CR or PR, according to the RECIST v.1.1 for target lesions and assessed by MRI: CR, complete response: Disappearance of all target lesions; PD, progressive disease: 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; PR, partial response: >=30% decrease in the sum of the longest diameter of target lesions; SD, stable disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; TF, treatment failure.
Time Frame: Minimum 10-12 months if negative results and up to 26-28 months if study is to be complete the targeted enrollment
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
Participants
  CR | 2 | 0 | 0
  PR | 20 | 1 | 3
  SD | 24 | 9 | 17
  PD | 8 | 10 | 13
  TF | 0 | 0 | 1

3. Secondary Outcome: Duration of Response
Description: Duration of response (DoR), defined as the time between the date when the response criteria (PR or CR, whichever was first reached) were fulfilled to the first date when disease progression (PD), recurrence or death was documented. According to the RECIST v.1.1 for target lesions and assessed by MRI: CR, complete response: Disappearance of all target lesions; PD, progressive disease: 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; PR, partial response: >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Minimum 10-12 months if negative results and up to 26-28 months if study is to be complete the targeted enrollment
Population: Responder patients (PR or CR, whichever was first reached)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 22 | 1 | 3
months | 6.3 [3.4 to 12.7] | 2.7 [NA to NA] — Only 1 patient | 3.6 [2.1 to 16.1]
Statistical Analysis 1: Comparison: Cohort A (BRCA+) vs Cohort A1 (BRCA+/PARPi) vs Cohort B (Unselected); Test type: Superiority; p = 0.0909, Log Rank

4. Secondary Outcome: Duration of Response Rate at 6 Months
Description: as for outcome 3
Time Frame: Time between the response criteria date and the date when disease progression, recurrence or death was documented, up to 6 months
Population: Responder patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 22 | 1 | 3
percentage of participants | 53.1 [31.8 to 74.4] | 0 [NA to NA] — Only 1 patient | 33.3 [0 to 86.7]

5. Secondary Outcome: Duration of Response Rate at 12 Months
Description: as for outcome 3
Time Frame: Time between the response criteria date and the date when disease progression, recurrence or death was documented, up to 12 months
Population: Responder patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 22 | 1 | 3
percentage of participants | 33.8 [13.5 to 54.1] | 0 [NA to NA] — Only 1 patient | 33.3 [0 to 86.7]

6. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit, defined as the percentage of patients with ORR or SD lasting over three months (SD >3 months).
  The overall response rate is defined as the percentage of patients with a confirmed response, either complete response (CR) or partial response (PR), according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1. Per RECIST v1.1 for target lesions and assessed by MRI: CR, Disappearance of all target lesions; PR >=30% decrease in the sum of the longest diameter of target lesions.
  SD, stable disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Minimum 10-12 months if negative results and up to 26-28 months if study is to be complete the targeted enrollment
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 61.1 [46.9 to 74.1] | 40.0 [19.1 to 63.9] | 32.4 [17.4 to 50.5]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the period of time from the date of first infusion to the date of progression disease, death (due to any cause), or last tumor evaluation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 36 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
months | 4.6 [3.0 to 6.2] | 1.4 [1.3 to 3.9] | 2.5 [1.3 to 3.4]
Statistical Analysis 1: Comparison: Cohort A (BRCA+) vs Cohort A1 (BRCA+/PARPi) vs Cohort B (Unselected); Test type: Superiority; p = 0.002, Log Rank

8. Secondary Outcome: Progression-free Survival at 3 Months
Description: Progression-free survival (PFS), defined as the period of time from the date of first infusion to the date of PD, death (due to any cause), or last tumor evaluation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from the date of first infusion to the date of PD, death (due to any cause), or last tumor evaluation, up to 3 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 63.5 [50.4 to 76.6] | 42.5 [20.3 to 64.7] | 35.5 [18.9 to 52.1]

9. Secondary Outcome: Progression-free Survival at 6 Months
Description: as for outcome 8
Time Frame: Time from the date of first infusion to the date of PD, death (due to any cause), or last tumor evaluation, up to 6 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 37.6 [24.2 to 50.9] | 21.3 [2.8 to 39.7] | 11.1 [0 to 22.6]

10. Secondary Outcome: Progression-free Survival at 12 Months
Description: as for outcome 8
Time Frame: Time from the date of first infusion to the date of PD, death (due to any cause), or last tumor evaluation, up to 12 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 20.5 [9.1 to 31.9] | 0 [0 to 0] | 3.7 [0 to 10.7]

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be defined as time from the date of first infusion to the date of death or last contact
Time Frame: 36 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
months | 18.6 [10.9 to 22.8] | 8.1 [4.6 to 14.6] | 12.1 [6.6 to 17.9]
Statistical Analysis 1: Comparison: Cohort A (BRCA+) vs Cohort A1 (BRCA+/PARPi) vs Cohort B (Unselected); Test type: Superiority; p = 0.0561, Log Rank

12. Secondary Outcome: Overall Survival Rate at 12 Months
Description: Overall survival (OS), defined as the time from the date of first infusion to the date of death or last contact
Time Frame: Time from the date of first infusion to the date of death or last contact, up to 12 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 62.5 [49.0 to 75.9] | 29.7 [7.9 to 51.5] | 55.4 [37.9 to 73.0]

13. Secondary Outcome: Overall Survival Rate at 18 Months
Description: Overall survival (OS), defined as the time from the date of first infusion to the date of death or last contact.
Time Frame: Time from the date of first infusion to the date of death or last contact, up to 18 months
Population: Cohort A: Two patients never treated; Cohort B: 1 patient due to lack of post-baseline tumor assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
Number analyzed (Participants) | 54 | 20 | 34
percentage of participants | 53.4 [39.2 to 67.5] | 22.3 [1.6 to 42.9] | 27.7 [11.5 to 43.9]

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, aproximately 6 years
Description: Two patients in Cohort A were never treated with lurbinectedin and therefore were not included in the analysis of safety
Arm/Group | Cohort A (BRCA+) | Cohort A1 (BRCA+/PARPi) | Cohort B (Unselected)
All-Cause Mortality (participants affected / at risk) | 40/54 | 13/20 | 30/35
Serious Adverse Events (participants affected / at risk) | 14/54 | 5/20 | 8/35
Other Adverse Events (participants affected / at risk) | 54/54 | 20/20 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (BRCA+) (N=54) | Cohort A1 (BRCA+/PARPi) (N=20) | Cohort B (Unselected) (N=35)
anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (9) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug interaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (4) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Listeriosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (BRCA+) (N=54) | Cohort A1 (BRCA+/PARPi) (N=20) | Cohort B (Unselected) (N=35)
anaemia (Blood and lymphatic system disorders) | 13 (16) | 2 (3) | 6 (10)
febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 24 (48) | 11 (15) | 7 (9)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 5 (8) | 1 (1) | 1 (1)
diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 11 (25) | 5 (6) | 7 (12)
constipation (Gastrointestinal disorders) | 23 (32) | 9 (17) | 9 (17)
diarrhoea (Gastrointestinal disorders) | 16 (23) | 4 (7) | 5 (6)
dyspepsia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3)
nausea (Gastrointestinal disorders) | 43 (123) | 15 (23) | 20 (37)
odynophagia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 23 (48) | 7 (9) | 10 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
chills (General disorders) | 1 (1) | 2 (2) | 1 (1)
fatigue (General disorders) | 48 (195) | 10 (21) | 30 (66)
Gait disturbance (General disorders) | 1 (3) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 3 (4) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 13 (15) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (4) | 0 (0)
Oedema (General disorders) | 5 (13) | 2 (2) | 4 (5)
pain (General disorders) | 3 (4) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 8 (10) | 4 (5) | 6 (16)
Chest discomfort (General disorders) | 0 (0) | 2 (3) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (9) | 1 (1) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Sputum purulent (Infections and infestations) | 0 (0) | 0 (0) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 24 (48) | 11 (15) | 7 (9)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 15 (20) | 6 (7) | 5 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (5) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 2 (2) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 7 (9) | 2 (3) | 3 (4)
Dysgeusia (Nervous system disorders) | 3 (8) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 16 (29) | 6 (10) | 5 (5)
Neuralgia (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 8 (9) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 2 (2) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 5 (11) | 8 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 1 (1) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Lymphoedema (Vascular disorders) | 4 (5) | 0 (0) | 4 (5)
Phlebitis (Vascular disorders) | 4 (5) | 2 (3) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review

DOCUMENTS (2):
  • Study Protocol (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT01525589/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT01525589/SAP_001.pdf